CLINICAL TRIAL: NCT05985902
Title: The Efficiency of Different Exercise Methods in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUsyildirim03
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic scoliosis; Schroth Exercises; Scoliosis Specific Exercises; Trunk Muscle Strength; Respiratory Muscle Strength; Muscle Stiffness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Core stabilization exercise training will be given to the control group for 12 weeks, 7 days a week, for 60 minutes. Core stabilization exercises will be applied to this group under the supervision of a physiotherapist for 2 days in our unit, while home-based core stabilization exercise training will be given on other days of the week.
  Interventions: Other: Core Stabilization Exercises
- Training Group (Experimental): After the first evaluation, the training group will be given Schroth exercise training for 12 weeks, 7 days a week, for 60 minutes. This group will be given Schroth exercises under the supervision of a physiotherapist for 2 days in our unit, while home-based Schroth exercise training will be given on other days of the week.
  Interventions: Other: Schroth Exercises

INTERVENTIONS:
Other: Core Stabilization Exercises — Core stabilization training; exercises for 2 muscle systems that contribute to spinal stability are given. The first one is the "local system" muscles; multifidus, transversus abdominis, diaphragm and pelvic floor muscles. The second, the "global system" includes large superficial muscles, such as erector spines, rectus abdominis, internal and external obliques, quadratus lumborum, gluteus ma
  Arms: Control Group
Other: Schroth Exercises — In the Schroth exercise training, there are 3-dimensional exercises that include the principles of axial reach, deflection, derotation, rotational breathing and stabilization.
  Arms: Training Group

SUMMARY:
The vertebral column is a structure that transfers the weight of the head and torso to the lower extremity, provides trunk movements and protects the spinal cord.A three dimensional deformity involving lateral flexion of the vertebrae in the frontal plane at 10 ° and above, including axial rotation and physiologic flexion (hypokyphosis) components in the sagittal plane, is defined as scoliosis. Adolescent idiopathic scoliosis (AIS) is a type of idiopathic scoliosis that occurs in the period from the onset of puberty (up to 10 years) until the closure of growth plates.

Scoliosis is caused by postural, balance and neuromotor disorders as a primary cause of impaired sensory integrity, proprioceptive feedback deficits, secondary lung problems, organ disorders and pain. In addition, the quality of life in these individuals is also seen to decrease.

There are no studies in the literature examining the effects of Schroth exercise training on trunk muscle strength, respiratory muscle strength, trunk muscle stiffness, balance and quality of life in children with adolescent idiopathic scoliosis.

The aim of our study is to examine whether Schroth exercise training has an effect on trunk muscle strength, trunk muscle stiffness, respiratory muscle strength, balance, quality of life and perception of cosmetic deformity in children with adolescent idiopathic scoliosis. It is thought that this study will fill the gap in the literature with the original information it will bring to the literature and will shed light on future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AIS scoliosis
* Individuals agreeing to participate in the study
* Patients between the ages of 10-20
* Patients with AIS whose Cobb angle measured on X-ray is between 15-40 degrees

Exclusion Criteria:

* Documented diagnosis any of cardiopulmonary, neurological, orthopedic or mental disorders which may affect the assessments results.
* Patients previously undertaken any of spinal surgeries.
* Patients involved in exercise training 3 or more days a week

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Isokinetic Muscle Strength | Baseline and after 12 weeks
  In order to examine the muscle strength of the patients and the effectiveness of the treatment, the muscle strength of the individuals will be evaluated with the Biodex System 3-Pro (Biodex Medical Systems, Inc, New York, USA) isokinetic dynamometer device. The Biodex isokinetic dynamometer device adapts at a constant speed, allowing a dynamic test that can give resistance. The adaptiveness of the resistance and the ability to give the same resistance throughout the entire range of motion provide maximum muscle strength. In addition to this situation, the performance of the muscles can be evaluated at different angular velocities. Muscle function and muscle strength can be determined during maximum muscle contraction by using a linear scale with isokinetic dynamometer, which is an objective assessment, and with this method, information about the strength of the upper and lower extremities and trunk muscles can be obtained.
Muscle Stiffness | Baseline and after 12 weeks
  Shear Wave Elastography, also known as dynamic elastography, is a sonoelastography examination that has been developed and rapidly developed in recent years, and it provides additional information about tissue properties by evaluating tissue flexibility that can contribute to the diagnosis. In this technique application, a short-term, high-power acoustic repulsive radiation force is applied to the tissue with ultrasound probes. This force causes small displacements in tissues. These displacements in the horizontal plane are called "shear waves" and the rate of progression of these waves in the tissue can be measured. The shear wave velocity is directly proportional to the hardness of the tissue. The velocity values obtained show the objective elasticity values. Patients' spinal and abdominal muscle stiffness will be evaluated with the Toshiba Aplio 500 (Toshiba Medical Systems Corporation, Japan).
Respiratory Muscle Strength | Baseline and after 12 weeks
  Respiratory muscle strength will be measured with a portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical; UK). Pressures will be assessed by measurements of maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) during a few seconds of maximal inspiration (Müller maneuver) and expiration (Valsalva maneuver) by mouth.
Postural Stability | Baseline and after 12 weeks
  Postural Stability and balance will be evaluated with the Biodex Balance System®. The Biodex Balance System® is a validated and reliable instrument used to assess postural stability, limits of stability and fall risk. It consists of balance platform, arm supports, screen and printer. The platform can be adjusted as static or mobile (12 levels of movement amount; level 12 is the most stable, level 1 is the least stable level that can move up to 20 degrees in each direction) according to the test to be applied.
Cobb Angle | Baseline and after 12 weeks
  The Cobb angle records at the first visit of the patients. The Cobb angle is the angle between the lines drawn perpendicular to the endplates first and last vertebrae involved in the curvature.
Angle of Trunk Rotation | Baseline and after 12 weeks
  Measurement will be applied with Bunnell Scoliometer by physiotherapist.
Quality of Life (Scoliosis Research Society-22) | Baseline and after 12 weeks
  Measurement will be applied with Scoliosis Research Society-22 Questionnaire. The scale consists of 22 questions and 5 subgroups of questions. Subgroups; pain, evaluation of general appearance, spinal functions, mental health and satisfaction with treatment. All of these sections can be evaluated separately and/or all questions can be evaluated by summing up under the total score. Scores are calculated by assigning an answer value to all 22 questions within a 5-point indicator chart. Each statement has responses ranging from negative to positive. The most negative answer; 1 and the most positive gets 5 points. High scores on the scale indicate an increase in quality of life, and low scores indicate a decrease.
Cosmetic Deformity Perception | Baseline and after 12 weeks
  Measurement will be applied with The Walter Reed Visual Assessment Scale. In the scale, deformity is categorized with 7 different aspects. Each of the 7 items contains a set of 5 figures representing the severity of the deformity. In these sets, there are visuals evaluating spine deformity, rib protrusion, waist protrusion, chest deformity, trunk imbalance, shoulder asymmetry and scapular asymmetry. The visuals include posterior views of the deformity and assess the patient's sense of how other people see their back. The selected images are scored as the lowest "1" and the highest "5", and the higher the total score obtained, the more negative-worse the perceived deformity is defined.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No